CLINICAL TRIAL: NCT03747744
Title: Phase I Clinical Trial on Intratumoral Injection of Autologous CD1c (BDCA-1)+ Myeloid Dendritic Cells Plus Talimogene Laherparepvec (T-VEC)
Brief Title: Intratumoral Injection of Autologous CD1c (BDCA-1)+ Myeloid Dendritic Cells Plus Talimogene Laherparepvec (T-VEC)
Acronym: myDCTV
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-BN-002
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec

STUDY DESIGN:
Intervention Model Description: Intratumoral injection of T-VEC followed by intratumoral injection of CD1c (BDCA-1)+ myDC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD1c (BDCA-1)+ myDC (Experimental): CD1c (BDCA-1)+ myDC
  Interventions: Other: CD1c (BDCA-1)+ myDC

INTERVENTIONS:
Other: CD1c (BDCA-1)+ myDC — Intratumoral injection in subcutaneous, cutaneous, soft tissue metastases
  Other Names: intratumoral injection of talimogene laherparepvec (T-VEC)

SUMMARY:
Over the past few years it has become evident that cancer cells can be recognized by the patient's own immune system. The immunological mechanisms at play are often referred to as the "cancer immune cycle" (Chen and Mellman 2013; Mellman 2013; Chen and Mellman 2017).In immune-evasive tumors a pivotal role has been attributed to myeloid dendritic cells (myDC) in regulating the activity of anti-tumor CTL activity within the TME (Broz, Binnewies et al. 2014). In animal models, myDC have been demonstrated to play an essential role in "licensing" anti-tumor CTLs to eradicate tumor cells. These myDC also migrate to tumor-draining lymph nodes and present tumor antigens to T-cells in these secondary lymphoid organs (Roberts, Broz et al. 2016). Human myDCs exist in two subsets that are differentiated by expression of either the BDCA-1 or BDCA-3 surface marker. The CD1c (BDCA-1)+ antigen is specifically expressed on human dendritic cells, which are CD11chighCD123low and represent the major subset of myDCs in human blood (about 0.6 % of all peripheral blood mononuclear cells (PBMCs)). CD1c (BDCA-1)+ myDC play an important role in the cross-presentation of tumor antigens following immunogenic cell death (Di Blasio, Wortel et al. 2016). Under conditions of tumor growth, myDC will be poorly recruited to the tumor microenvironment, do not get activated and thereby fail to efficiently coordinate anti-tumor immunity within the tumor micro-environment and present tumor associated antigens within tumor-draining lymph nodes. Talimogene laherparepvec (T-VEC) is a first-in-class oncolytic virus based on a modified herpes simplex virus (HSV) type 1 designed to selectively replicate in and lyse tumor cells while promoting regional and systemic antitumor immunity. In this phase I clinical trial we propose to investigate the safety of intratumoral injection of autologous CD1c (BDCA-1)+ myDC in non-visceral metastases of melanoma plus intratumoral injection of T-VEC (at its approved dose and regimen for the treatment of melanoma). We hypothesize that CD1c (BDCA-1)+ myDC in the T-VEC inflamed tumor microenvironment of the metastasis will capture tumor antigens in vivo and through cross-presentation of these antigens coordinate an effective anti-tumor T-cell response.

DETAILED DESCRIPTION:
Over the past few years it has become evident that cancer cells can be recognized by the patient's own immune system. The immunological mechanisms at play are often referred to as the "cancer immune cycle" (Chen and Mellman 2013; Mellman 2013; Chen and Mellman 2017). Remarkable anti-tumor activity has been achieved by blocking the inhibitory T-cell receptor CTLA-4 and/or the PD-1/-L1 axis. Immune checkpoint inhibition by monoclonal antibody (mAb) therapy has become a standard of care in patients with advanced melanoma, renal cell carcinoma, non-small cell lung carcinoma, Hodgkin's lymphoma and bladder cancer. Indications are still expanding. Activity of PD-1 and CTLA-4 inhibition has been correlated with hallmarks of pre-existing anti-tumor T-cell response (e.g. presence of cytotoxic T lymphocytes (CTL) in the tumor microenvironment (TME), PD-L1 expression in response to T-cell secreted IFN-gamma and transcriptional evidence for CTL-activity), mutational load of the cancer cells and presence of highly immunogenic neo-epitopes in the cancer cell genome (Tumeh, Harview et al. 2014). In immune-evasive tumors a pivotal role has been attributed to myeloid dendritic cells (myDC) in regulating the activity of anti-tumor CTL activity within the TME (Broz, Binnewies et al. 2014). In animal models, myDC have been demonstrated to play an essential role in "licensing" anti-tumor CTLs to eradicate tumor cells. Activation of oncogenic signaling pathways such as the WNT/beta-Catenin pathway can lead to the exclusion of myeloid DC's from the TMZ (Spranger, Bao et al. 2015; Spranger and Gajewski 2016). Absence of myDCs at the invasive margin and within metastases has been correlated with defective CTL activation allowing the metastasis to escape the anti-tumor immune response (Salmon, Idoyaga et al. 2016). These myDC also migrate to tumor-draining lymph nodes and present tumor antigens to T-cells in these secondary lymphoid organs (Roberts, Broz et al. 2016). Presence of myeloid DC's was more strongly correlated with T-cell infiltration into tumors as compared to neo-antigen load in 266 melanomas from The Cancer Genome Atlas(Spranger, Luke et al. 2016). Human myDCs exist in two subsets that are differentiated by expression of either the BDCA-1 or BDCA-3 surface marker. The CD1c (BDCA-1)+ antigen is specifically expressed on human dendritic cells, which are CD11chighCD123low and represent the major subset of myDCs in human blood (about 0.6 % of all peripheral blood mononuclear cells (PBMC)). CD1c (BDCA-1)+ myDC have a monocytoid morphology and express myeloid markers such as CD13 and CD33 as well as Fc receptors such as CD32, CD64, and FceRI. Furthermore, myDC are determined to be CD4+, Lin (CD3, CD16, CD19, CD20, CD56)-, CD2+, CD45RO+, CD141 (BDCA-3)-low, CD303 (BDCA-2)-, and CD304 (BDCA-4/Neuropilin-1)-. A proportion of CD1c (BDCA-1)+ myDC co-expresses CD14 and CD11b. These dual positive cells for CD14+ and CD1c (BDCA-1) have immunosuppressive capacity and inhibit T-cell proliferation in vitro. Depletion of this cell type is preferred prior to using CD1c (BDCA-1)+ cells for immunostimulatory purposes (Bakdash, Buschow et al. 2016; Schroder, Melum et al. 2016). CD1c (BDCA-1)+ myDC play an important role in the cross-presentation of tumor antigens following immunogenic cell death (Di Blasio, Wortel et al. 2016). Under conditions of tumor growth, myDC will be poorly recruited to the tumor microenvironment, do not get activated and thereby fail to efficiently coordinate anti-tumor immunity within the tumor micro-environment and present tumor associated antigens within tumor-draining lymph nodes. When activated appropriately, human CD1c (BDCA-1)+ dendritic cells secrete high levels of IL-12 and potently prime CTL responses (Nizzoli, Krietsch et al. 2013). In vitro, IL-12 production by CD1c (BDCA-1)+ myDC can be boosted by exogenous IFN-gamma. (Nizzoli, Krietsch et al. 2013) CD1c (BDCA-1)+ myDC spontaneously "partially mature" within 12 hours following their isolation. Optimal maturation with secretion of IFN-gamma as well as the orientation of stimulated T-lymphocytes towards a Th1 phenotype is only achieved following Toll-like receptor stimulation.(Skold, van Beek et al. 2015) Talimogene laherparepvec (T-VEC; Imlygic) is a first-in-class oncolytic virus based on a modified herpes simplex virus (HSV) type 1 designed to selectively replicate in and lyse tumor cells while promoting regional and systemic antitumor immunity. T-VEC is modified through the deletion of two nonessential viral genes. Functional deletion of the herpes virus neurovirulence factor gene (ICP34.5) attenuates viral pathogenicity and enhances tumor-selective replication. T-VEC is further modified by deletion of the ICP47 gene to reduce virally mediated suppression of antigen presentation and increase the expression of the HSV US11 gene. Insertion and expression of the gene encoding human granulocyte macrophage colony-stimulating factor (GM-CSF) results in local GM-CSF production to recruit and activate antigen presenting cells with subsequent induction of tumor-specific T cell responses. T-VEC has been evaluated in early-phase studies, which demonstrated intratumoral replication and expression of GM-CSF and an acceptable safety profile (low-grade fever, chills, myalgias, and injection site reactions) after intralesional administration. In a single arm phase II study, an overall response rate (ORR) of 26% was reported in patients with stage IIIc to IV melanoma, with responses observed in both injected and non-injected lesions, including visceral lesions. Biopsy of regressing lesions suggested an association between response and presence of IFN- producing MART-1-specific CD8+ T cells and reduction in CD4+ FoxP3+ regulatory T cells, consistent with induction of host antitumor immunity. The efficacy and toxicity of T-VEC in advanced melanoma was evaluated in a randomized phase III trial comparing intratumoral T-VEC injections with subcutaneous GM-CSF injections. With T-VEC, the primary end point of durable response rate (DRR; continuous response lasting > 6 months) was significantly higher (16% vs 2%; odds ratio, 8.9; P,.001), ORR improved (26% vs 6%), and the overall survival (OS) improved numerically but not statistically by 4.4 months (hazard ratio, 0.79; 95% CI, 0.62 to 1.00; P = .051). Tumor regression was seen in tumors both injected and not injected with T-VEC. The incidence of grade 3/4 T-VEC-related adverse events (AEs) was 11%. (Andtbacka, Kaufman et al. 2015) In an open-label, multicenter, phase Ib trial, the combination of T-VEC with ipilimumab had a tolerable safety profile, and the combination appeared to have greater efficacy than either T-VEC or ipilimumab monotherapy.(Puzanov, Milhem et al. 2016) The combination of T-VEC plus pembrolizumab (an anti-PD1 monoclonal antibody) was associated with clinical benefit in advanced melanoma, as assessed by ORR and CR rate (Ribas, Dummer et al. 2017). A randomized, double-blind phase 3 trial of T-VEC plus pembrolizumab vs T-VEC placebo plus pembrolizumab is ongoing. In this phase I clinical trial we propose to investigate the safety of intratumoral injection of autologous CD1c (BDCA-1)+ myDC in non-visceral metastases of melanoma plus intratumoral injection of T-VEC (at its approved dose and regimen for the treatment of melanoma).

We hypothesize that CD1c (BDCA-1)+ myDC in the T-VEC inflamed tumor microenvironment of the metastasis will capture tumor antigens in vivo and through cross-presentation of these antigens coordinate an effective anti-tumor T-cell response.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures.
* Male or female age ≥ 18 years at the time of informed consent
* All subjects must have histologically confirmed advanced melanoma that cannot be completely surgically resected and have failed all standard curative and live prolonging therapy.
* All subjects must have non-visceral metastatic disease localizations that are amenable to intra-tumor injection by clinical and ultrasound (US) guidance. These metastases should be amenable to a safe post-injection biopsy (partial or complete).
* ECOG performance status of 0 or 1
* Candidate for intralesional therapy defined as either one of the following: a) at least 1 injectable cutaneous, subcutaneous, or nodal melanoma lesion ≥ 10 mm in longest diameter, b) multiple injectable melanoma lesions that in aggregate have a longest diameter of ≥ 10 mm injectable disease
* Adequate organ function determined within 28 days prior to enrollment, defined as follows: a) Hematological, i) Absolute neutrophil count ≥ 1500/mm3 (1.5x109/L) ii) Platelet count: ≥ 75.000/mm3 (7.5x109/L) iii) Hemoglobin: ≥ 8 g/dL (without need for hematopoietic growth factor or transfusion support) b) Renal, i) Serum creatinine: 1.5 x upper limit of normal (ULN), OR 24-hour creatinine clearance ≥ 60 mL/min for subject with creatinine levels > 1.5 x ULN. (Note: Creatinine clearance need not be determined if the baseline serum creatinine is within normal limits. Creatinine clearance should be calculated per institutional standard). c) Hepatic, i) Serum bilirubin: 1.5 x ULN OR direct bilirubin ≤ ULN for a subject with total bilirubin level > 1.5 x ULN ii) Aspartate aminotransferase (AST): 2.5 x ULN OR ≤ 5 x ULN for subject with liver metastases iii) Alanine aminotransferase (ALT): 2.5 x ULN OR ≤ 5 x ULN for subject with liver metastases d) Coagulation, i) International normalization ratio (INR) or prothrombin time (PT): 1.5 x ULN unless the subject is receiving anticoagulant therapy as long as PT and partial thromboplastin time (PTT)/ activated PTT (aPTT) is within therapeutic range of intended use of anticoagulants ii) PTT or aPTT: 1.5 x ULN unless the subject is receiving anticoagulant therapy as long as PT and PTT/aPTT is within therapeutic range of intended use of
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Subject has a tumor sample (archival sample obtained within 3 months prior to study participation or newly obtained biopsy). Subject must submit the tumor sample during screening. Subjects with a non-evaluable archival sample may obtain a new biopsy and subjects with a non-evaluable newly obtained biopsy may undergo re-biopsy at the discretion of the investigator.
* Adequate vascular access to undergo a leucapheresis.

Exclusion Criteria:

* Known active central nervous system (CNS) metastases. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids >10 mg/day of prednisone or equivalent. The exception does not include carcinomatosus meningitis which is excluded regardless of clinical stability.
* History or evidence of active autoimmune disease that requires systemic treatment (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History or evidence of melanoma associated with immunodeficiency states (e.g., hereditary immune deficiency, organ transplant, or leukemia)
* History of other malignancy within the past 5 years with the following exceptions: i) Malignancy treated with curative intent and with no known active disease present and has not received chemotherapy for > 5 years before enrollment and felt to be at low risk for recurrence by the treating physician ii) Adequately treated non-melanoma skin cancer without evidence of disease at the time of enrollment iii) Adequately treated cervical carcinoma in situ without evidence of disease at the time of enrollment iv) Adequately treated breast ductal carcinoma in situ without evidence of disease at the time of enrollment v) Prostatic intraepithelial neoplasia without evidence of prostate cancer at the time of enrollment vi) Adequately treated superficial or in-situ carcinoma of the bladder without evidence of disease at the time of enrollment
* Prior therapy with T-VEC or any other oncolytic viruses
* Prior treatment of other tumor vaccine
* Receive live vaccine within 28 days prior to enrollment
* Prior chemotherapy, radiotherapy, biological cancer therapy, targeted therapy, or major surgery within 28 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to enrollment.
* Currently receiving treatment in another investigational device or drug study, or less than 28 days since ending treatment on another investigational device or drug study
* Expected to require other cancer therapy while on study with the exception of local radiation treatment to the site of bone and other metastasis for palliative pain management
* Other investigational procedures while participating in this study are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | through study completion, up to 1 year
  Safety of intratumoral injection with CD1c (BDCA-1)+ myDC and intratumoral injection of T-VEC

CONTACTS AND LOCATIONS:
Overall Officials: Bart Neyns, MD,PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwarze JK, Tijtgat J, Awada G, Cras L, Vasaturo A, Bagnall C, Forsyth R, Dufait I, Tuyaerts S, Van Riet I, Neyns B. Intratumoral administration of CD1c (BDCA-1)+ and CD141 (BDCA-3)+ myeloid dendritic cells in combination with talimogene laherparepvec in immune checkpoint blockade refractory advanced melanoma patients: a phase I clinical trial. J Immunother Cancer. 2022 Sep;10(9):e005141. doi: 10.1136/jitc-2022-005141. PMID 36113895